### Title: Efficacy of a Health Belief Model Based Intervention for Anticoagulation Adherence

NCT number: NCT03864900

Document date:2017.4.20

### **Study Protocol**

**BACKGROUND**: Inconsistent anticoagulation therapy in AF patients is associated with a higher risk of stroke and abnormal bleeding. However, control of oral anticoagulation therapy in AF patients has been frequently reported as inadequate. Few theoretical based interventions have been tested for enhancing medication adherence in this population. Previous studies showed that the health belief model may offer some advantage over other behavior change theories for enhancing medication adherence in adult with chronic conditions.

**PURPOSE**: The purpose of the study is to investigate the efficacy of a health belief model based self-management of oral anticoagulant therapy intervention on the outcome of medication adherence and the mediators of knowledge, professional support, health belief, and self-efficacy in patients treated with oral anticoagulants for atrial fibrillation.

METHODS: The study is a randomized clinical trial with repeated measurements. A convenient sample of 72 adults who were treated with anticoagulants for atrial fibrillation was recruited from two teaching hospitals in northern Taiwan. Participants were randomly assigned 1:1 to either the control group (n = 36) or the intervention group (n = 36) after completion of baseline questionnaires. Allocation was balanced by site by using a minimization method. The health belief model based selfmanagement intervention comprised two main components: a 60-minute individual face-to-face instruction and six follow-up telephone calls. Participants in the control group received regular medication education, 10-minute individual instruction for health knowledge and six follow-up telephone calls for concerning health. Data were collected at baseline, third month, and sixth month in both groups, by using self-administered questionnaires. The investigator administered the study questionnaire after obtaining informed consent from each subject. The data collection took place at the waiting areas outside the outpatient clinics during the patients' visits to the clinics. For subjects who were unable to read the questionnaire due to vision or other problems, the investigator read each question to help them complete the questionnaire. The instruments include the Atrial Fibrillation Knowledge Scale, Satisfaction Scale about Service and Warfarin Treatment, Belief about Anticoagulation Survey, and Self-Efficacy for Appropriate Medication Use Scale.

DATA ANALYSIS: Data were analyzed using the Statistical Package for Social Sciences 20.0 (SPSS, Inc., Chicago, IL, USA). Descriptive analyses were used to describe study variables. Independent t-tests and one-way analysis of variance (ANOVA) were performed to analyze the baseline equivalent between study groups. The generalized estimating equations were used to analyze the efficacy of the intervention for enhancing knowledge, knowledge, perceived benefits, perceived barriers, self-efficacy, and adherence to anticoagulant therapies in patients treated with oral anticoagulants for atrial fibrillation.

### ClinicalTrials.gov

A service of the National Institutes of Health

### Participant Flow Data Preparation Checklist

**Overview:** The Participant Flow module is a tabular summary of participants' progress through each stage of a study by assignment group. Use this checklist with the <u>Participant Flow Template</u> and <u>Results Data Element Definitions</u> to complete this module of the results section.

| Select | Information to have available for Participant Flow | Data Element |
|---|---|---|
| | <ul> <li>Conceptual overview of the study design, including the type (e.g., single group, cross-over, parallel) and any distinct stages (e.g., double-blind then open-label)</li> <li><u>Tip</u>: Have a <u>CONSORT flow diagram</u> available.</li> </ul> | |
| | <ul> <li>Description of any significant study events that occurred after participants were<br/>enrolled, but before they were assigned to a study group (e.g., run-in phase or<br/>washout)</li> </ul> | [*]Pre-assignment<br>Details |
| ⊠ | <ul> <li>Number of groups that accurately describes the study design from participant assignment to completion</li> <li><u>Tip</u>: The number of groups is typically equal to the number of unique paths (participant experiences) in a CONSORT flow diagram, from beginning to end. Each group will be reported as a table column.</li> </ul> | *Arm/Group<br>Information |
| | <ul> <li>For each group: <ul> <li>Title—Descriptive label for the group</li> <li><u>Tip</u>: Use informative labels (e.g., "Placebo"), not generic labels (e.g., "Group 1"). The label will become the header for that table column.</li> <li>Description—Detailed explanation of the interventions administered or the groups observed during each stage of the study</li> <li><u>Tip</u>: Include details about the intervention (e.g., dosage, dosage form, frequency and duration of administration) or observation.</li> </ul> </li> </ul> | *Arm/Group<br>Title<br>*§Arm/Group<br>Description |
| | Number of discrete stages or intervals of activity in the study | *Period(s) |
| | <ul> <li>Descriptive title for each period (the default for one Period is "Overall Study")</li> <li>Tip: A Period Title should describe what happened during that period of the study. For example, "Double-blind (0 to 24 weeks)" and "Open-label (24 to 48 weeks)" are more descriptive than "Period 1" and "Period 2."</li> </ul> | *Period Title |
| | <ul> <li>Number of participants that Started and Completed each period:</li> <li>Started—Participants initiating each period (e.g., the number of participants assigned or randomized to each group for that period)</li> <li><u>Tip</u>: If the number of participants starting the first period is different from the total enrolled in the study, explain why in Pre-assignment Details.</li> <li>Completed—Participants still in the study at the end of the period</li> <li><u>Tip</u>: If the unit of assignment is a unit other than participants, specify the name of the unit (e.g., eyes, lesions, implants) and provide the number of units.</li> <li><u>Tip</u>: Each unit of assignment (participants or units other than participants) should only be represented in one group. For example, if the unit of assignment is participants, do not count a participant more than once by including them in more than one group.</li> <li><u>Tip</u>: Use the Additional Milestone field to record any specific events or time points in the study between the Started and Completed milestones.</li> </ul> | *Started *Completed [*]Type of Units Assigned Additional Milestone |

'Required

\*§ Required if Primary Completion Date is on or after January 18, 2017
[\*] Conditionally required

## Participant Flow Template

| | [*] Pre-assignment Details |
|---|---|
| investigators to determine their eligibility | |
| porthern Taiwan. Potential participants were referred by cardiologists and screened by one of the | n |
| Patients with AFib were recruited from the cardiology clinics of two general hospitals in | Recruitment Details P |

### Period (1)

| [*] Other | [*] Other | | | | | | | | | | | | [*] Milestone | [*] Milestone | [*] Milestone | | | | | * | ( |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| [*] Other Operation | [*] other Change Medication | [*] Withdrawal by | [*] Protocol | [*] Pregnancy | [*] Physician | [*] Lost to | [*] Lack of Efficacy | [*] Death | [*] Adverse Event | | Not Completed | * Completed | | | | * Started | | *§ Arm/Group | * | Overall Study | |
| 1 | 1 | 1 | | | | | | | | Reason Not Completed Type ③ | | 33 | | | | 36 | Number of Participants (4) | Intervention Group | EG | 1 | |
| 0 | 2 | 2 | | | | | | | | Type ③ | (automatically calculated) | 30 | | | | 36 | Number of Participants (4) | Control Group | CG | | |
| | | | | | | | | | | | | | | | | | Number of Participants | | | | |

| Baseline Chara | Baseline Characteristics Template | | Age* (use | (use at least one) | one) | Clinic | Clinical Irials.gov | gov |
|---|---|---|---|---|---|---|---|---|
| | * Arm/Group Title | EG | | CG | | 01 | Total | |
| * | *§ Arm/Group Description ① | Intervention group | group | Control Group | Group | | | |
| * Overall Number | * Overall Number of Baseline Participants (2) | 36 | | 36 | | | | w |
| [*] Baseline Ana | [*] Baseline Analysis Population Description | Age 20 years and | over, | diagnosis with £ | AFib by a physica | physican and receving anticoagulation therapy | pagulation th | erapy |
| Age, Categorical | | | | | | | | |
| | <=18 years | 0 | | 0 | | | | (3) |
| | Between 18 and 65 years | 13 | | 13 | | | | ω |
| | >=65 years | 41 | | 42 | | | | (S) |
| * Unit of Measure | Participants | | | | | | | |
| Age, Continuous | | | | | | | | |
| * Measure Type | * Measure of Dispersion | | | | | | | |
| (Select One) Mean Median Least Squares Mean (LSM) | (Select One) Standard Deviation Inter-quartile Range Full Range | | | | | | | |
| Geometric LSM * Unit of Measure | years old | 69.3 | 7.5 | 73.3 | 10 | | _ | |
| Age, Customized | | | | | | | | |
| * Measure Type | * Measure of Dispersion | | | | | | | |
| (Select One) Count of Participants (4) Mean Median Least Squares Mean (LSM) Geometric Mean Geometric LSM Number Count of Units (4) | (Select One) Not Applicable (5) Standard Deviation Inter-Quartile Range Full Range | | | | | | | |
| [*] Row/Category Title (6) | | | 45 | | 45 | 49 | (3) | 45 |
| [*] Row/Category Title (6) | | | 4 5 | | 45 | 45 | 3 | 45 |
| * Unit of Measure | | | | | | | | |

<sup>\*§</sup> Required it Primary Completion Date is on or after January 18, 2017

Arm/Group Description describes details about the intervention strategy (e.g., dose, dosage form, frequency, duration) or groups evaluated.

Overall Number of Units Analyzed and Type of Units Analyzed may also be specified.

Total values are automatically calculated for Overall Number of Baseline Participants and for data reported with a Measure Type of Number, Count of Participants, or Count of Units.

<sup>\*</sup>Required
Arm/G
Overal
Total v
H Mea
G Not Ap
G Optio If Measure Type is a "count," percentage of participants/units is automatically calculated from Overall Number of Baseline Participants/Units Analyzed. The percentage can be hidden (display is optional).

<sup>[</sup>Optional] Add as many Rows/Categories as needed. If more than one is entered, a Row/Category Title and Baseline Measure Data are required for each row. Not Applicable should be used only if Measure Type is Number, Count of Participants, or Count of Units. No dispersion value is needed if Measure of Dispersion is Not Applicable.

**Baseline Characteristics Template** 

Sex/Gender\* (use at least one)

ClinicalTrials.gov

| *\$ Arm/Group Description ① * Overall Number of Baseline Participants ② [*] Baseline Analysis Population Description Sex: Female, Male * Unit of Measure * Unit of Measure * Unit of Measure * Measure Type (Select One) Count of Participants ④ Mean Mean Mean Mean Geometric LSM Number Count of Units ④ [*] Row/Category Title ⑥ [*] Row/Category Title ⑥ [*] Row/Category Title ⑥ |
|---|
| eline Participants |
| ysis Population Descripti |
| Fema |
| M |
| _ |
| nder, Customized |
| Row/Category Title ⑥ |
| Row/Category Title (6) |
| Row/Category Title ⑥ |
| * Unit of Measure |

<sup>&#</sup>x27;S Required it Primary Completion Date is oil of after January 10, 2011

Arm/Group Description describes details about the intervention strategy (e.g., dose, dosage form, frequency, duration) or groups evaluated.

Overall Number of Units Analyzed and Type of Units Analyzed may also be specified.

If Measure Type is a "count," percentage of participants/units is automatically calculated from Overall Number of Baseline Participants/Units Analyzed. The percentage can be hidden Total values are automatically calculated for Overall Number of Baseline Participants and for data reported with a Measure Type of Number, Count of Participants, or Count of Units.

<sup>60(5)</sup> Not Applicable should be used only if Measure Type is Number, Count of Participants, or Count of Units. No dispersion value is needed if Measure of Dispersion is Not Applicable. (display is optional)

<sup>[</sup>Optional] Add as many Rows/Categories as needed. If more than one is entered, a Row/Category Title and Baseline Measure Data are required for each row.

| <b>Baseline Characteristics Template</b> | plate Race*s, | s, Ethnicity*s, and Region | Cunical Irials. gov |
|---|---|---|---|
| * Arm/Group Title | EG | CG | Total |
| *§ Arm/Group Description ① | Intervention Group | Control Group | |
| * Overall Number of Baseline Participants ② | 36 | 36 | 72 |
| [*] Baseline Analysis Population Description | | | |
| Race (NIH/OMB) ④ | | | |
| American Indian or Alaska Native | | | |
| Asian | 36 | 36 | 72 |
| Native Hawaiian or Pacific Islander | | | |
| Black or African American | | | |
| White | | | |
| More than one race | | | |
| Unknown or Not Reported | | | |
| * Unit of Measure Participants | | | |
| Ethnicity (NIH/OMB) ④ | | | |
| Hispanic or Latino | | | |
| Not Hispanic or Latino | | | |
| Unknown or Not Reported | | | |
| * Unit of Measure Participants | | | |
| Region of Enrollment | | | |
| United States | | | |
| Region/Country Name (5) Taiwan | 36 | 36 | |
| Region/Country Name (5) | | | |
| Region/Country Name (5) | | | |
| * | | | |

<sup>\*§</sup> Required it Primary Completion Date is on or after January 18, 2017

Arm/Group Description describes details about the intervention strategy (e.g., dose, dosage form, frequency, duration) or groups evaluated.

Overall Number of Units Analyzed and Type of Units Analyzed may also be specified.

Total values are automatically calculated for Overall Number of Baseline Participants and for each Baseline Measure.

If not using NIH/OMB categories, use Race/Ethnicity, Customized (not shown); if not collected, use Race and Ethnicity Not Collected (not shown). [Optional] Region of Enrollment Baseline Measure is optional, but at least one Region/Country is required if reporting Region of Enrollment. Add as many Regions/Countries as needed.

### [\*] Row/Category Title 6 [\*] Row/Category Title 6 Least Squares Mean (LSM) Count of Participants (4) Baseline Characteristics Template Count of Units (4) Geometric Mean \* Measure Type Geometric LSM (Select One) \* Overall Number of Baseline Participants (2) \* Unit of Measure [\*] Baseline Analysis Population Description Number Median Mean [\*] Study-Specific Baseline Measure Title \*§ Arm/Group Description (1) **Baseline Measure Description** \* Measure of Dispersion Disease duration Inter-Quartile Range Standard Deviation Not Applicable (5) (Select One) \* Arm/Group Title Full Range month Intervention Group 65.6 History of anticoagulation therapy Patients with AFib currently receving anticoagulation therapy EG 45 Study-Specific Measure\*\$ 49(5) 4)(5) 70.9 Control Group 36 CG 66.2**4**5 49(5) **4**) (5) 49(5) ClinicalTrials.gov Total (2) (u) **495 4 5** (3)

<sup>\*§</sup> Required if Primary Completion Date is on or after January 18, 2017

<sup>[\*]</sup> Conditionally required

Arm/Group Description describes details about the intervention strategy (e.g., dose, dosage form, frequency, duration) or groups evaluated

Overall Number of Units Analyzed and Type of Units Analyzed may also be specified.

Total values are automatically calculated for Overall Number of Baseline Participants and for data reported with a Measure Type of Number, Count of Participants, or Count of Units.

If Measure Type is a "count," percentage of participants/units is automatically calculated from Overall Number of Baseline Participants/Units Analyzed. The percentage can be hidden (display

Not Applicable should be used only if Measure Type is Number, Count of Participants, or Count of Units. No dispersion value is needed if Measure of Dispersion is Not Applicable

<sup>(</sup>p)(v) required if more than one row [Optional] Add as many Rows/Categories as needed. If more than one is entered, a Row/Category Title and Baseline Measure Data are required for each row. Row/Category Titles are only

# Outcome Measure Template

| | | | | Ups to 24 weeks | * Outcome Measure Time |
|---|---|---|---|---|---|
| | | | adherence when taking anticoagulants | adherence whe | Description |
| ticipants' medicatio | Medications Scale (ARMS) assess the participants' medication | | adherence. The study adapted Adherence to Refills | adherence. The | [*] Outcome Measure |
| | | CCKS, illess is also seen a si p | C 1110111101 101 ab 10 17 11 | Lai ricibalità Mei | |
| or for medication | Anticoagulant medication adherence | reaks. These is the soons of o | Anticoagulant medication adherence | Anticoagulant m | * Outcome Measure |
| Post-Hoc | Other Pre-specified | Secondary | Primary | (Select One) | * Outcome Measure |

More details available in the Results Data Element Definitions. April 2017

| * Unit of | [*] Row/Category Title | [*] Row/Category Title | Least Squares Mean | Median | Mean | Count of Participants (3) | (Select One) | * Measure Type | | * | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| score | | Medication adherence | Inter-Quartile Range | Standard Error | Standard deviation | Not Applicable (4) | (Select One) | * Measure of | [*] Analysis Population | Number of Participants Analyzed | *§ Arm/Group Description | * Arm/Group |
| | | 8.1 | | | | | | | All participants with baseline and | 36 | Intervent | EG |
| | 34 | 1.4 | | | | | | | with baseline | 6 | Intervention group | G |
| | | 9.2 | | | | | | | at least fellow | w | Control group | ) |
| | 34 | 2.2 | | | | | | | at least fellow up for 24 weeks | 36 | group | CG |
| - 116 | 3.4 | 34 | | | | | | | | | | |

| Statisticat | Charles III |
|-------------|-------------|
| Analysis | 1 |
| iempiate | Theretain |

## ClinicalTrials.gov

| Other Statistical Analysis (4) | | | | | Method of<br>Estimation | | | of Hypothesis - | Statistical Test | | | Analysis<br>Overview | Statistical |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Estimation Comments (2) | Parameter Dispersion | Confidence Interval<br>(if applicable) | Estimated Value | [*] Estimation Parameter<br>(if applicable) | Comments (2) | [*] Method<br>(required if p-value entered) | Comments ② | [*] P-Value (if applicable) | [*] Comments ③ | * Type of Statistical Test | Comments ② | * Comparison Group Selection ① |
| A generalized estimating equation (GEE) 28 was used to model each outcome variable as a function of group effect, time effect, and group by time interaction effect. | | Type: (Select One) Standard Deviation Standard Error of the Mean Value: | Level: 95 % Confidence Interval Number of Sides: (Select One) Lower Limit: Upper Limit: Lower Limit: | 0.5 (calculated value) | (Select One) Cox Proportional Hazard Mean Difference (Net) Odds Ratio, Log Slope Hazard Ratio (HR) Median Difference (Final Values) Risk Difference (RD) Other Hazard Ratio, Log Median Difference (Net) Risk Ratio (RR) (generalized estimating equation) Mean Difference (Final Values) Odds Ratio (OR) Risk Ratio, Log | | (Select One) ANCOVA Fisher Exact Mixed Models Analysis t-Test, 1-Sided ANOVA Kruskal-Wallis Regression, Cox t-Test, 2-Sided Chi-Squared Log Rank Regression, Linear Wilcoxon Chi-Squared, Corrected Mantel Haenszel Regression, Logistic (Mann-Whitney) Cochran-Mantel-Haenszel McNemar Sign Test Other () | | 0.05 (calculated value, not the a priori threshold for statistical significance) | | (Select One) Superiority Equivalence Non-inferiority Other (for example, single group or other descriptive analysis) | | □ ✓Arm/Group1 □ ✓Arm/Group2 □ Arm/Group3 |

<sup>[\*]</sup> Conditionally required

Use the checkboxes to select the Arms/Groups (pre-populated from the Outcome Measure) involved in the statistical analysis.
 (2) (Optional) Include any relevant information about the row above (e.g., the null hypothesis, details of the power calculation, adjustment for multiple comparisons, the a priori threshold for statistical significance, the direction of the comparison). Do not include written results or conclusions.

<sup>(3)</sup> If a non-inferiority or equivalence analysis, information on the definition of the non-inferiority or equivalence margin is required.
(4) If the statistical analysis cannot be submitted using the Statistical Test of Hypothesis or Method of Estimation options, provide a description and the results

# All-Cause Mortality and Serious Adverse Events Template ClinicalTrials.gov

| [*] Adverse I<br>Source Vocabulary | *§ Time Frame [*] Adverse Event Reporting Description Source Vocabulary Name for Table Default ① | non | non applicable | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| *§ Collection Ap | *§ Collection Approach for Table Default ① | (Select One) | Systematic | atic | Non-Systematic | Lic . | | | 11 |
| × | Arm Coom Description (2) | | | | | | | | |
| *8 | *§ Arm/Group Description (2) | | | | | | | | ni. |
| *§ All-Cause Mortality | * | | | | | | | | |
| | | *§ Number<br>Participants<br>Affected | | *§ Number<br>Participants<br>at Risk | *§ Number Participants Affected | | *§ Number<br>Participants<br>at Risk | *§ Number<br>Participants<br>Affected | er |
| | *§ Total | | | | | | | | 1 |
| * Serious Adverse Events | ents | | | | | | | | 1 |
| | | * Number<br>Participants<br>Affected | * Number<br>Participants<br>at Risk | Number<br>Events | * Number<br>Participants<br>Affected | * Number<br>Participants<br>at Risk | Number<br>Events | * Number Participants Affected | * Number<br>Participants<br>at Risk |
| | * Total | | | | | | | | |
| * Adverse Event<br>Term | * Organ System | | | | | | | | |
| | 3 | | (4)[*] | | | <b>4</b> [*] | | | |
| | 3 | | <b>4</b> [*] | | | (4)[*] | | | |
| | (3) | | <b>4</b> [*] | | | <b>4</b> [*] | | | |
| | (3) | | <b>4</b> [*] | | | (4)[*] | | | T |
| | 3 | | (4)[*] | | | 4[*] | | | |
| | (3) | | <b>(</b> 4)[*] | | | <b>4</b> [*] | | | |

Required

<sup>\*§</sup> Required if Primary Completion Date is on or after January 18, 2017

<sup>[\*]</sup> Conditionally required

<sup>1)</sup> If entered, the table default values apply to all Adverse Event Terms. The values may be changed for any single Adverse Event, if different from the table default.
2) Arm/Group Description describes details about the intervention strategy (e.g., dose, dosage form, frequency, duration) or groups evaluated.
3) Organ System must be selected from a pick-list of high-level categories. See the Results Data Element Definitions for details.
4) Number of Participants at Risk for an Adverse Event Term is only required when the value differs from the Total Number of Participants at Risk.

# Other (Not Including Serious) Adverse Events Template

ClinicalTrials.gov

| | | | | | | | | | * Adverse Event<br>Term | | * Freque<br>Reporti | * Other (Not Including Serious) Adverse Events | | | *§ Collection / | | Source Vocabula | [*] Advers | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 20 | | | | | | | | | * Organ System | | * Frequency Threshold for<br>Reporting Other Adverse<br>Events (0–5%) | ding Serious) Adve | *§ Arm/Group Description ② | * Arm/( | *§ Collection Approach for Table Default (1) | | Source Vocabulary Name for Table Default ① | [*] Adverse Event Reporting Description | *§ T |
| | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | tem | * Total | % | rse Events | cription (2) | Arm/Group Title | Detault (1) | | Default ① | escription | *§ Time Frame |
| 7 | | | | | | | | | | | * Number<br>Participants<br>Affected | | | | (select One) | 75-12 | | | non aı |
| Africal Indian | <b>(</b> 4)[*] | <b>(4)[*]</b> | (4)[*] | <b>(</b> 4)[*] | <b>(4)[*]</b> | (*) | (4)[*] | <b>4</b> [*] | | | * Number<br>Participants<br>at Risk | | | | J SYSTEILIALIC | | | | non applicable |
| 210 2017 | | | | | | | | | | | Number<br>Events | | | | שנוכ | <del>+</del> . | | | |
| [*] | | | | | | | | | | | * Number<br>Participants<br>Affected | | | | NOH-3ystematic | Non Customat | | | |
| (*) Conditionally required | <b>4</b> [*] | 4[*] | <b>4</b> [*] | <b>4</b> [*] | 4[*] | <b>4</b> [*] | <b>4</b> [*] | <b>4</b> [*] | | | * Number<br>Participants<br>at Risk | 0 | | | <del>.</del> | 5 | | | |
| required | | | | | | | | | | | Number<br>Events | | | | | | | | |
| | | | | | | | | | | | * Number Participants Affected | | | | | | | | |
| | (4)[*] | (4)[*] | <b>4</b> [*] | 4[*] | 4[*] | <b>4</b> [*] | <b>(4)[*]</b> | <b>(4)[*]</b> | | | * Number Participants at Risk | | | | | | | | |
| | | | | | | | | | | | Number<br>Events | | | | | | | | |

Kequirea

<sup>3</sup> Required if Primary Comple

If entered, the table default values apply to all Adverse Event Terms. The values may be changed for any single Adverse Event, if different from the table default.
 Arm/Group Description describes details about the intervention strategy (e.g., dose, dosage form, frequency, duration) or groups evaluated.
 Organ System must be selected from a pick-list of high-level categories. See the Results Data Element Definitions for details.
 Number of Participants at Risk for an Adverse Event Term is only required when the value differs from the Total Number of Participants at Risk.